CLINICAL TRIAL: NCT03382834
Title: Selective Estrogen Receptor Modulators to Enhance the Efficacy of Viral Reactivation With Histone Deacetylase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5366; 38190 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2019-12-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Tamoxifen; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Tamoxifen + Vorinostat (Experimental): From Day 0 to Day 38, participants will receive tamoxifen orally once a day. On Days 35 and 38, participants will receive a single dose of vorinostat orally.
  Interventions: Drug: Tamoxifen; Drug: Vorinostat; Drug: Antiretroviral drugs
- Arm B: Vorinostat alone (Active Comparator): Day 0 to Day 38 will be an observation period with no tamoxifen. On Days 35 and 38, participants will receive a single dose of vorinostat orally.
  Interventions: Drug: Vorinostat; Drug: Antiretroviral drugs

INTERVENTIONS:
Drug: Tamoxifen — 20 mg orally
  Arms: Arm A: Tamoxifen + Vorinostat
Drug: Vorinostat — 400 mg orally
Drug: Antiretroviral drugs — Participants will receive antiretroviral drugs provided by their own doctors. Antiretroviral drugs will not be provided by the study.

SUMMARY:
This study evaluated the effects of tamoxifen exposure in combination with vorinostat on viral reactivation among HIV-1 infected post-menopausal women with virologic suppression on antiretroviral therapy (ART), when compared to vorinostat alone.

DETAILED DESCRIPTION:
The selective estrogen receptor modulator (SERM) tamoxifen may enhance the ability of the histone deacetylase inhibitor (HDACi) vorinostat to reverse HIV-1 latency. This study evaluated the safety of tamoxifen therapy combined with vorinostat and the effectiveness of this combination on latent virus reactivation in HIV-1 infected post-menopausal women with virologic suppression on antiretroviral therapy, when compared to vorinostat alone.

The study was conducted in two steps. During Step 1, the study enrolled women with HIV into two groups. Arm A received tamoxifen daily for 38 days, plus a single dose of vorinostat on Days 35 and 38. Arm B had a 38-day observation period with no tamoxifen, plus a single dose of vorinostat on Days 35 and 38. All participants continued to take ART drugs prescribed by their doctors. ART drugs were not be provided by the study.

Study visits during Step 1 occurred at Days 0, 28, 35, 38, 45, and 65. Study visits could include physical examinations, blood collection, electrocardiograms, and adherence assessments.

During Step 2, all participants were followed for 240 additional weeks for annual long-term safety follow-up. These visits were conducted by phone and collected information from participants on vital status and any new cancer diagnoses.

Step 1 and Step 2 have been completed and this results submission pertains to both.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Postmenopausal at study entry with agreement not to participate in assisted reproductive technology in the future.
* CD4+ cell count greater than 300 cells/uL obtained within 90 days prior to study entry.
* Continuous antiretroviral therapy (ART) for at least 2 years prior to enrollment with no known interruption in therapy for greater than 7 days within 90 days prior to study entry.
* Plasma HIV-1 RNA level of less than 20 copies/mL obtained by Roche HIV-1 viral load assay or less than 40 copies/mL obtained by the Abbott assay, within 90 days prior to study entry.
* Ability and willingness of potential participant to provide written informed consent.

Exclusion Criteria:

* History of venous thromboembolism.
* History of stroke.
* Known history of hypercoagulable state.
* Tobacco smoking or e-cigarette use within 90 days prior to study entry.
* History of any malignancy requiring systemic chemotherapy or systemic immunotherapy.
* History of endometrial or breast cancer or known genetic testing with BRCA positive results indicating an increased risk for breast and ovarian cancer.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, or investigational therapy within 60 days prior to study entry.
* Any systemic hormonal therapy defined as oral or injectable contraceptives, estrogen and combined estrogen-progesterone replacement therapy in the prior 12 months, or a hormone containing intrauterine device (IUD) within 6 months prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gandhi, MD, Study Chair — Massachusetts General Hospital (MGH) CRS; Eileen Scully, MD, PhD, Study Chair — Johns Hopkins University
Locations (15):
- United States (14):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by the NIH.
Access Criteria: With whom?
  Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  For what types of analyses?
  To achieve aims in the proposal approved by the AIDS Clinical Trials Group. By what mechanism will data be made available?
  Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data."

REFERENCES:
- [Derived] Scully EP, Aga E, Tsibris A, Archin N, Starr K, Ma Q, Morse GD, Squires KE, Howell BJ, Wu G, Hosey L, Sieg SF, Ehui L, Giguel F, Coxen K, Dobrowolski C, Gandhi M, Deeks S, Chomont N, Connick E, Godfrey C, Karn J, Kuritzkes DR, Bosch RJ, Gandhi RT. Impact of Tamoxifen on Vorinostat-Induced Human Immunodeficiency Virus Expression in Women on Antiretroviral Therapy: AIDS Clinical Trials Group A5366, The MOXIE Trial. Clin Infect Dis. 2022 Oct 12;75(8):1389-1396. doi: 10.1093/cid/ciac136. PMID 35176755
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables

RESULTS

PARTICIPANT FLOW:
Period: Step 1
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Started | 21 | 10
Completed (Completed Step 1 of the study.) | 21 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Step 2
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Started | 21 | 9
Completed | 17 | 7
Not Completed | 4 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Site Terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [54 to 61] | 55 [51 to 59] | 57 [53 to 60]
Age, Customized [Count of Participants; unit: Participants]
  Age categorized: < 50 years | 2 | 1 | 3
  Age categorized: 50 - 59 years | 11 | 7 | 18
  Age categorized: >= 60 years | 8 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 17 | 8 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 9 | 3 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 1 | 0 | 1
  United States | 20 | 10 | 30
Baseline Cell-associated HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/million CD4 cells] — Baseline cell-associated HIV-1 RNA levels (CA-RNA) (log10 copies/mL) were measured in CD4 T-cells. Baseline CA-RNA was calculated as the average of the pre-entry and entry CA-RNA results. Population: CA-RNA analyses were performed on the efficacy population, defined as the subset of enrolled participants who received full study treatment and did not have ART interruption or confirmed viral load (VL) >= 200 copies/mL. The definition was expanded by team to exclude 2 participants; one with high pre-entry VL and one with wrong timing of samples.
  log10 copies/million CD4 cells
    number analyzed (Participants) | 19 | 8 | 27
    (all) | 1.81 [1.38 to 2.49] | 2.5 [2.01 to 3.15] | 2.17 [1.56 to 2.69]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With New Grade 3 or Greater Adverse Events
Description: Proportion of participants with new Grade 3 or greater adverse events that are considered definitely, probably, or possibly related to study treatment (as judged by the core protocol team). The DAIDS AE Grading Table (corrected Version 2.1, July 2017) was used.
Time Frame: Measured from study entry through Day 65
Population: Enrolled participants who were exposed to study treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Number analyzed (Participants) | 21 | 9
proportion of participants | 0 [0 to 0.13] | 0 [0 to 0.28]

2. Primary Outcome: Change From Baseline in Cell-associated HIV-1 RNA in CD4+ T Cells
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value of Cell-associated HIV-1 RNA on Day 38 (5 hours post vorinostat) minus the value at baseline.
Time Frame: Pre-entry, entry, and Day 38
Population: Efficacy population
Measure: Mean (95% Confidence Interval); unit: log10 copies/million CD4 cells
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Number analyzed (Participants) | 19 | 8
log10 copies/million CD4 cells | 0.06 [-0.24 to 0.36] | 0.17 [-0.15 to 0.50]
Statistical Analysis 1: Comparison: Arm A: Tamoxifen + Vorinostat vs Arm B: Vorinostat Alone; Test type: Superiority; p = 0.68, t-test, 1 sided; The hypothesis was that tamoxifen would enhance the HIV transcription effect of vorinostat (i.e., log10 change would be greater in Arm A than Arm B)

3. Secondary Outcome: Number of Participants With HIV-1 RNA Levels (Measured by Single Copy Assay) Greater or Equal to the Lower Limit of Quantification
Description: Number of participants with HIV-1 RNA levels measured by single copy assay (SCA) greater or equal to the lower limit of quantification (LOQ). The lower limit of quantification for this study was 0.47 copies/mL.
Time Frame: Pre-entry, entry, Day 28, Day 35, Day 38 (5 hours post vorinostat), Day 45, Day 65
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Number analyzed (Participants) | 19 | 8
Participants
  Pre-entry SCA >= LOQ | 10 | 6
  Entry SCA >=LOQ | 9 | 3
  Day 28 SCA >=LOQ | 11 | 4
  Day 35 SCA >=LOQ | 11 | 5
  Day 38 SCA >=LOQ | 7 | 5
  Day 45 SCA >=LOQ | 9 | 4
  Day 65 SCA >=LOQ | 10 | 5

4. Secondary Outcome: Change From Baseline in Total HIV-1 DNA Levels in CD4+ T Cells
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value of Total HIV-1 DNA on Day 38 (5 hours post vorinostat) minus the value at baseline.
Time Frame: Pre-entry, entry, and Day 38
Population: Efficacy Population
Measure: Mean (95% Confidence Interval); unit: log10 copies/million CD4 cells
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
Number analyzed (Participants) | 19 | 8
log10 copies/million CD4 cells | 0 [-0.12 to 0.13] | -0.04 [-0.33 to 0.25]
Statistical Analysis 1: Comparison: Arm A: Tamoxifen + Vorinostat vs Arm B: Vorinostat Alone; Test type: Superiority; p = 0.73, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From study entry to end of study
Description: The protocol required reporting of all diagnoses, all signs/symptoms/laboratory values Grade ≥ 3, and all diagnoses/signs/symptoms/laboratory values that led to treatment change or met SAE or EAE reporting requirements through Day 65 (Step 1), and all new cancer diagnoses/deaths during the subsequent 240 week long-term safety follow-up (Step 2). For grading, sites referred to the Division of AIDS AE Grading Table, corrected Version 2.1, July 2017.
Arm/Group | Arm A: Tamoxifen + Vorinostat | Arm B: Vorinostat Alone
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 3/21 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Tamoxifen + Vorinostat (N=21) | Arm B: Vorinostat Alone (N=10)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03382834/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03382834/SAP_000.pdf